CLINICAL TRIAL: NCT00005140
Title: Epidemiology of Cardiovascular and Non-Cardiovascular Risk In Chicago
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1011; R01HL021010 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease; Cerebrovascular Disorders; Diabetes Mellitus; Hypertension; Cerebrovascular Accident
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease; Cerebrovascular Disorders; Diabetes Mellitus; Hypertension; Stroke

SUMMARY:
To continue the comprehensive research program on the epidemiology of cardiovascular and other major chronic diseases, including cancer and diabetes, in four Chicago population cohorts. The four cohorts include the Chicago Heart Association Detection Project in Industry cohort, the Peoples Gas Company cohort first examined in 1958-1959, the Peoples Gas Company cohort first examined in 1959-1962, and the Western Electric Company cohort.

DETAILED DESCRIPTION:
BACKGROUND:

Over the last forty years, epidemiologic studies have made basic contributions to knowledge of the etiology and natural history of the chronic diseases -- cardiovascular diseases, diabetes, and cancers. Findings from the epidemiologic studies have provided practical foundations for the development of prevention and control programs to improve life styles and to control high blood pressure by drugs, when indicated. These developments and their impact on life styles and risk factors have probably contributed to the marked decline in mortality rates from coronary heart disease, stroke, all cardiovascular disease, and all causes throughout the 1970s and 1980s.

The four epidemiologic studies have as their foundation the major contributions of the earlier 'first generation' epidemiological studies including the Albany Civil Servant Study, the Charleston Study, the Framingham Heart Study, the Tecumseh Study and others. The significance of these studies lies in their potential for elucidating key 'second generation' issues in the epidemiology of the major cardiovascular and non-cardiovascular chronic diseases.

DESIGN NARRATIVE:

Chicago Heart Association Detection Project in Industry: Employees of 85 firms in the greater Chicago area were screened between the Fall of 1967 to early 1973. The total labor force among these companies was over 75,000 persons. The volunteer rate for the screening was 55 percent. All employees were encouraged to participate irrespective of job type or shift worked. At each employment site data were collected on smoking habits, previous medical diagnosis, current treatments for hypertension, heart disease and diabetes, height and weight, age, sex, race, heart rate.

Peoples Gas Company: All data on the two cohorts were collected as part of the periodic medical examination program for all employees in the Medical Department of the Company by its full-time staff of physicians. Data were collected on age, race, height, weight, blood pressure, serum cholesterol, smoking history, heart rate, resting ECG, medical and family history, alcohol and coffee and tea consumption, education, military service, occupation, physical activity, diet, and glucose and serum uric acid levels. Repeat exams were scheduled yearly for men 50-59, every two years for men 40-49, and every four years for men 25-39.

Western Electric Company: This longitudinal study of coronary heart disease was initiated in 1957 at the Hawthorne Works of the Western Electric Company in Chicago. The male subjects were free of coronary heart disease at baseline. The medical history and physical examination were modeled after the Framingham Heart Study. Data were collected on diet, physical activity, electrocardiogram, blood hemoglobin and blood cholesterol levels, body fatness, blood pressure, height, weight, lipoprotein lipase, glucose level, and smoking.

The study was renewed in FY 1992 and again in FY 1998. The 1998 renewal used data and analyses from the four cohorts. It focused on six specific aims: factors influencing coronary heart disease-cardiovascular disease risk long-term in young adult women and men (ages 18 to 39 at baseline); factors influencing coronary heart disease-cardiovascular disease risk long-term in African-American women and men; factors influencing coronary heart disease-cardiovascular disease risk during both earlier and later follow-up (first 15 years and beyond 15 years of follow-up); impact of baseline low risk status on long-term risk of mortality from coronary heart disease, cardiovascular disease, non-cardiovascular disease, and all causes; relationship of habitual intake of multiple food groups to 10 year change in serum cholesterol, blood pressure, weight, and to 30-year risks of death from coronary heart disease, cardiovascular disease, cancers, and all causes; differences in risk factors impact between groups based on sex, race, age, or risk factor status.

The study has been extended through July 2005 and uses data and analyses from the Chicago Heart Association Detection Project in Industry cohort. The study focuses on three specific aims: factors influencing coronary heart disease and cardiovascular disease risk long-term in young adult women (ages 18-39 at baseline); factors influencing coronary heart disease and cardiovascular disease risk long-term in young adult and middle-aged African American men and women; and the impact of baseline "low risk" status on long-term mortality from coronary heart disease, cardiovascular disease, non-cardiovascular disease, and all causes in young adult women (ages 18-39), including African-American and white women.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1977-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Greenland — Northwestern University

REFERENCES:
- [Background] LeGrady D, Dyer AR, Shekelle RB, Stamler J, Liu K, Paul O, Lepper M, Shryock AM. Coffee consumption and mortality in the Chicago Western Electric Company Study. Am J Epidemiol. 1987 Nov;126(5):803-12. doi: 10.1093/oxfordjournals.aje.a114717. PMID 3661528
- [Background] Liao Y, Liu K, Dyer A, Schoenberger JA, Shekelle RB, Collette P, Stamler J. Sex differential in the relationship of electrocardiographic ST-T abnormalities to risk of coronary death: 11.5 year follow-up findings of the Chicago Heart Association Detection Project in Industry. Circulation. 1987 Feb;75(2):347-52. doi: 10.1161/01.cir.75.2.347. PMID 3492312
- [Background] Liu K. Measurement error and its impact on partial correlation and multiple linear regression analyses. Am J Epidemiol. 1988 Apr;127(4):864-74. doi: 10.1093/oxfordjournals.aje.a114870. PMID 3354551
- [Background] Clay CM, Dyer AR, Liu K, Stamler J, Shekelle RB, Berkson DM, Paul O, Schoenberger JA, Lepper M, Lindberg HA, et al. Education, smoking and non-cardiovascular mortality: findings in three Chicago epidemiological studies. Int J Epidemiol. 1988 Jun;17(2):341-7. doi: 10.1093/ije/17.2.341. PMID 3403129
- [Background] Levine W, Dyer AR, Shekelle RB, Schoenberger JA, Stamler J. Serum uric acid and 11.5-year mortality of middle-aged women: findings of the Chicago Heart Association Detection Project in Industry. J Clin Epidemiol. 1989;42(3):257-67. doi: 10.1016/0895-4356(89)90061-9. PMID 2709083
- [Background] Levine W, Dyer AR, Shekelle RB, Schoenberger JA, Stamler J. Post-load plasma glucose and cancer mortality in middle-aged men and women. 12-year follow-up findings of the Chicago Heart Association Detection Project in Industry. Am J Epidemiol. 1990 Feb;131(2):254-62. doi: 10.1093/oxfordjournals.aje.a115495. PMID 2296978
- [Background] Dyer AR, Stamler J, Shekelle RB. Serum cholesterol and mortality from coronary heart disease in young, middle-aged, and older men and women from three Chicago epidemiologic studies. Ann Epidemiol. 1992 Jan-Mar;2(1-2):51-7. doi: 10.1016/1047-2797(92)90037-q. PMID 1342265
- [Background] Vaccaro O, Ruth KJ, Stamler J. Relationship of postload plasma glucose to mortality with 19-yr follow-up. Comparison of one versus two plasma glucose measurements in the Chicago Peoples Gas Company Study. Diabetes Care. 1992 Oct;15(10):1328-34. doi: 10.2337/diacare.15.10.1328. PMID 1425098
- [Background] Shekelle RB, Tangney CC, Rossof AH, Stamler J. Serum cholesterol, beta-carotene, and risk of lung cancer. Epidemiology. 1992 Jul;3(4):282-7. doi: 10.1097/00001648-199207000-00003. PMID 1637892
- [Background] Goff DC Jr, Shekelle RB, Katan MB, Gotto AM Jr, Stamler J. Does body fatness modify the association between dietary cholesterol and risk of coronary death? Results from the Chicago Western Electric Study. Arterioscler Thromb. 1992 Jul;12(7):755-61. doi: 10.1161/01.atv.12.7.755. PMID 1616901
- [Background] Stamler J. Diet and coronary heart disease. Biometrics. 1982 Mar;38 Suppl:95-118. PMID 7046825
- [Background] Liu K, Stamler J, Stamler R, Cooper R, Shekelle RB, Schoenberger JA, Berkson DM, Lindberg HA, Marquardt J, Stevens E, Tokich T. Methodological problems in characterizing an individual's plasma glucose level. J Chronic Dis. 1982;35(6):475-85. doi: 10.1016/0021-9681(82)90062-5. PMID 7076788
- [Background] Circulating cholesterol level and risk of death from cancer in men aged 40 to 69 years. Experience of an international collaborative group. JAMA. 1982 Dec 3;248(21):2853-9. doi: 10.1001/jama.1982.03330210035031. PMID 7143647
- [Background] Liu K, Cedres LB, Stamler J, Dyer A, Stamler R, Nanas S, Berkson DM, Paul O, Lepper M, Lindberg HA, Marquardt J, Stevens E, Schoenberger JA, Shekelle RB, Collette P, Shekelle S, Garside D. Relationship of education to major risk factors and death from coronary heart disease, cardiovascular diseases and all causes, Findings of three Chicago epidemiologic studies. Circulation. 1982 Dec;66(6):1308-14. doi: 10.1161/01.cir.66.6.1308. No abstract available. PMID 6814786
- [Background] Dyer AR, Stamler J, Shekelle RB, Schoenberger JA, Stamler R, Shekelle S, Berkson DM, Paul O, Lepper MH, Lindberg HA. Relative weight and blood pressure in four Chicago epidemiologic studies. J Chronic Dis. 1982;35(12):897-908. doi: 10.1016/0021-9681(82)90121-7. PMID 7174772
- [Background] Larbi EB, Cooper RS, Stamler J. Alcohol and hypertension. Arch Intern Med. 1983 Jan;143(1):28-9. No abstract available. PMID 6849605
- [Background] Stamler J. Nutrition-related risk factors for the atherosclerotic diseases--present status. Prog Biochem Pharmacol. 1983;19:245-308. No abstract available. PMID 6338524
- [Background] Trevisan M, Ostrow D, Cooper R, Liu K, Sparks S, Okonek A, Stevens E, Marquardt J, Stamler J. Abnormal red blood cell ion transport and hypertension. The People's Gas Company study. Hypertension. 1983 May-Jun;5(3):363-7. doi: 10.1161/01.hyp.5.3.363. PMID 6840823
- [Background] Stamler J, Stamler R, Liu K: High Blood Pressure: Role in Coronay Heart Disease, and Implications for Prevention and Control. In: Connor WE, Bristow DJ (Eds), Coronary Heart Disease - Prevention, Complications, and Treatment, Lippincott, Philadelphia, Pa, p 85-109, 1985
- [Background] Stamler J, Farinaro E, Riccardi G, Stamler R, Mancini M: Does asymptomatic Hyperglycemia Always Have to be Treated? (Italian), J Ital Diabetol, 3:1-7, 1983
- [Background] Trevisan M, Tsong Y, Stamler J, Tokich T, Mojonnier L, Hall Y, Cooper R, Moss D. Nervous tension and serum cholesterol: findings from the Chicago Coronary Prevention Evaluation Program. J Human Stress. 1983 Mar;9(1):12-6. doi: 10.1080/0097840X.1983.9935020. PMID 6886402
- [Background] Stamler J. The prevention and control of epidemic coronary heart disease: scientific foundations and strategic approaches. Int J Cardiol. 1983 Sep;4(2):207-15. doi: 10.1016/0167-5273(83)90138-9. No abstract available. PMID 6629535
- [Background] Kaplan NM, Stamler J (Eds): Prevention of Coronary Heart Disease--Practical Management of the Risk Factors, WB Saunders, Philadelphia, 1983
- [Background] Stamler J, Liu K: The Benefits of Prevention. In: Kaplan NM, Stamler J (Eds), Prevention of Coronary Heart Disease--Practical Management of the Risk Factors, WB Saunders, Philadelphia, pp 188-207, 1983
- [Background] Stamler R, Stamler J: 'Mild' Hypertension: Risks and Strategy. Parts I and II. Primary Cardiol, 9(10):150-166, Oct, and 9(11):12-25, Nov, 1983
- [Background] Stamler J, Stamler R, Liu K: High Blood Pressure: Role in Coronary Heart Disease, and Implications for Prevention and Control. Position Paper Prepared at the Request of the Non-Communicable Disease Division, and the Cardiovascular Section, World Health Organization, Geneva, Switzerland, WHO/CVD/83.5, 8th August, 1983
- [Background] Stamler J: Does Cholesterol Change Alter Coronary Artery Disease Risk? Epidemiological Evidence. Proceedings of a Symposium on the Decline in Coronary Heart Disease Mortality--the Role of Cholesterol Change. Science and Medicine, New York, pp 27-45, 1983
- [Background] Coffee and cholesterol. N Engl J Med. 1983 Nov 17;309(20):1248-50. doi: 10.1056/NEJM198311173092012. No abstract available. PMID 6633576
- [Background] Ueshima H, Cooper R, Stamler J, Yu C, Tatara K, Asakura S. Age specific mortality trends in the U.S.A. from 1960 to 1980: divergent age-sex-color patterns. J Chronic Dis. 1984;37(6):425-39. doi: 10.1016/0021-9681(84)90026-2. PMID 6725497
- [Background] Kannel WB, Doyle JT, Ostfeld AM, Jenkins CD, Kuller L, Podell RN, Stamler J. Optimal resources for primary prevention of atherosclerotic diseases. Atherosclerosis Study Group. Circulation. 1984 Jul;70(1):155A-205A. PMID 6327117
- [Background] Larbi EB, Stamler J, Dyer A, Cooper R, Paul O, Shekelle RB, Lepper M. The population attributable risk of hypertension from heavy alcohol consumption. Public Health Rep. 1984 May-Jun;99(3):316-9. PMID 6429732
- [Background] Cooper R, Liu K, Stamler J, Schoenberger JA, Shekelle RB, Collette P, Shekelle S. Prevalence of diabetes/hyperglycemia and associated cardiovascular risk factors in blacks and whites: Chicago Heart Association Detection Project in Industry. Am Heart J. 1984 Sep;108(3 Pt 2):827-33. doi: 10.1016/0002-8703(84)90678-1. PMID 6475752
- [Background] Trevisan M, Ostrow D, Cooper RS, Sempos C, Stamler J. Sex and race differences in sodium-lithium countertransport and red cell sodium concentration. Am J Epidemiol. 1984 Oct;120(4):537-41. doi: 10.1093/oxfordjournals.aje.a113914. PMID 6475923
- [Background] Stamler J: The Prevention of Coronary Heart Disease (CHD). 1. Scientific Foundations--Recent Data. European Conference on Primary Prevention of Coronary Heart Disease, Anacapri, 15-19 October 1984. World Health Organization, Geneva, Switzerland. ICP/NCD 001/15, 15 October 1984
- [Background] Cooper R, Trevisan M, Ostrow D, Sempos C, Stamler J. Blood pressure and sodium-lithium countertransport: findings in population-based surveys. J Hypertens. 1984 Oct;2(5):467-71. doi: 10.1097/00004872-198410000-00004. PMID 6530551
- [Background] Stamler J: The Central and Essential Role of Nutrition in the Primary and Secondary Prevention of Coronary Heart Disease and Hypertension. In: Lovenberg W, Yamori Y, (Eds), Nutritional Prevention of Cardiovascular Disease, Academic Press, New York, NY, pp 383-405, 1984
- [Background] Stamler J, Stamler R, Liu K: High Blood Pressure. In: Connor WE, Bristow D (Eds), Coronary Heart Disease--Prevention, Complications, and Treatment, JB Lippincott, Philadelphia, Pa, pp 85-109, 1985
- [Background] Giumetti D, Liu K, Stamler R, Schoenberger JA, Shekelle RB, Stamler J. Need to prevent and control high-normal and high blood pressure, particularly so-called "mild" hypertension: epidemiological and clinical data. Prev Med. 1985 Jul;14(4):396-412. doi: 10.1016/0091-7435(85)90002-7. PMID 3877923
- [Background] Stamler R. Influence of treatment of "mild" hypertension on coronary heart disease. Acta Med Scand Suppl. 1985;701:89-99. doi: 10.1111/j.0954-6820.1985.tb08894.x. PMID 3907299
- [Background] Pan WH, Cedres LB, Liu K, Dyer A, Schoenberger JA, Shekelle RB, Stamler R, Smith D, Collette P, Stamler J. Relationship of clinical diabetes and asymptomatic hyperglycemia to risk of coronary heart disease mortality in men and women. Am J Epidemiol. 1986 Mar;123(3):504-16. doi: 10.1093/oxfordjournals.aje.a114266. PMID 3946397
- [Background] Dyer AR. A method for combining results from several prospective epidemiologic studies. Stat Med. 1986 Jul-Aug;5(4):303-17. doi: 10.1002/sim.4780050403. PMID 3764222
- [Background] Fish consumption and mortality from coronary heart disease. N Engl J Med. 1985 Sep 26;313(13):820-4. doi: 10.1056/NEJM198509263131311. No abstract available. PMID 4033711
- [Background] Liao YL, Emidy LA, Dyer A, Hewitt JS, Shekelle RB, Paul O, Prineas R, Stamler J. Characteristics and prognosis of incomplete right bundle branch block: an epidemiologic study. J Am Coll Cardiol. 1986 Mar;7(3):492-9. doi: 10.1016/s0735-1097(86)80458-2. PMID 3950228
- [Background] Nanas S, Pan WH, Stamler J, Liu K, Dyer A, Stamler R, Schoenberger JA, Shekelle RB. The role of relative weight in the positive association between age and serum cholesterol in men and women. J Chronic Dis. 1987;40(9):887-92. doi: 10.1016/0021-9681(87)90189-5. PMID 3496349
- [Background] Pan WH, Nanas S, Dyer A, Liu K, McDonald A, Schoenberger JA, Shekelle RB, Stamler R, Stamler J. The role of weight in the positive association between age and blood pressure. Am J Epidemiol. 1986 Oct;124(4):612-23. doi: 10.1093/oxfordjournals.aje.a114434. PMID 3489410
- [Background] Persky V, Pan WH, Stamler J, Dyer A, Levy P. Time trends in the US racial difference in hypertension. Am J Epidemiol. 1986 Nov;124(5):724-37. doi: 10.1093/oxfordjournals.aje.a114448. PMID 3766506
- [Background] Stamler J, Giumetti D, Liu K, Stamler R, Dyer A: The Risks of Hypertension. Proceedings of the Symposium on Control of Arterial Hypertension in the Prevention of Cardiovascular Disease, Hohenreid, Federal Republic of Germany, 1986.
- [Background] Liu K. Statistical issues related to the design of dietary survey methodology for NHANES III. Vital Health Stat 4. 1992 Mar;(27):3-14; discussion 15-23. No abstract available. PMID 1375411
- [Background] Crews DE, Stamler J, Dyer A. Conditions other than underlying cause of death listed on death certificates provide additional useful information for epidemiologic research. Epidemiology. 1991 Jul;2(4):271-5. doi: 10.1097/00001648-199107000-00006. PMID 1912042
- [Background] Almada SJ, Zonderman AB, Shekelle RB, Dyer AR, Daviglus ML, Costa PT Jr, Stamler J. Neuroticism and cynicism and risk of death in middle-aged men: the Western Electric Study. Psychosom Med. 1991 Mar-Apr;53(2):165-75. doi: 10.1097/00006842-199103000-00006. PMID 2031070
- [Background] Persky V, Ostrow D, Langenberg P, Ruby E, Bresolin L, Stamler J. Hypertension and sodium transport in 390 healthy adults in Chicago. J Hypertens. 1990 Feb;8(2):121-8. doi: 10.1097/00004872-199002000-00005. PMID 2162874
- [Background] Orencia AJ, Daviglus ML, Dyer AR, Shekelle RB, Stamler J. Fish consumption and stroke in men. 30-year findings of the Chicago Western Electric Study. Stroke. 1996 Feb;27(2):204-9. doi: 10.1161/01.str.27.2.204. PMID 8571410
- [Background] Gann PH, Daviglus ML, Dyer AR, Stamler J. Heart rate and prostate cancer mortality: results of a prospective analysis. Cancer Epidemiol Biomarkers Prev. 1995 Sep;4(6):611-6. PMID 8547827
- [Background] Pandey DK, Shekelle R, Selwyn BJ, Tangney C, Stamler J. Dietary vitamin C and beta-carotene and risk of death in middle-aged men. The Western Electric Study. Am J Epidemiol. 1995 Dec 15;142(12):1269-78. doi: 10.1093/oxfordjournals.aje.a117594. PMID 7503047
- [Background] Xie X, Liu K, Stamler J, Stamler R. Ethnic differences in electrocardiographic left ventricular hypertrophy in young and middle-aged employed American men. Am J Cardiol. 1994 Mar 15;73(8):564-7. doi: 10.1016/0002-9149(94)90334-4. PMID 8147301
- [Background] Stamler J, Dyer AR, Shekelle RB, Neaton J, Stamler R. Relationship of baseline major risk factors to coronary and all-cause mortality, and to longevity: findings from long-term follow-up of Chicago cohorts. Cardiology. 1993;82(2-3):191-222. doi: 10.1159/000175868. PMID 8324780
- [Background] Birmingham B, Dyer AR, Shekelle RB, Stamler J. Subscapular and triceps skinfold thicknesses, body mass index and cardiovascular risk factors in a cohort of middle-aged employed men. J Clin Epidemiol. 1993 Mar;46(3):289-302. doi: 10.1016/0895-4356(93)90077-e. PMID 8455054
- [Background] Goff DC Jr, Shekelle RB, Moye LA, Katan MB, Gotto AM Jr, Stamler J. Does body fatness modify the effect of dietary cholesterol on serum cholesterol? Results from the Chicago Western Electric Study. Am J Epidemiol. 1993 Jan 15;137(2):171-7. doi: 10.1093/oxfordjournals.aje.a116657. PMID 8452121
- [Background] Stamler J. The mass treatment of hypertensive disease: defining the problem. Ann N Y Acad Sci. 1978 Mar 30;304:333-62. doi: 10.1111/j.1749-6632.1978.tb25611.x. No abstract available. PMID 360924
- [Background] Stamler J. Hypertension, blood lipids, and cigarette smoking as co-risk factors for coronary heart disease: discussion. Ann N Y Acad Sci. 1978 Mar 30;304:140-6. doi: 10.1111/j.1749-6632.1978.tb25586.x. No abstract available. PMID 280227
- [Background] Stamler J. George Lyman Duff Memorial Lecture. Lifestyles, major risk factors, proof and public policy. Circulation. 1978 Jul;58(1):3-19. doi: 10.1161/01.cir.58.1.3. PMID 348343
- [Background] Stamler R, Stamler J. Where do we go in hypertension screening? Urban Health. 1978 Jun;7(5):8-9, 16. No abstract available. PMID 10308605
- [Background] Stamler J: Improving Life Styles to Control the Coronary Epidemic. Proceedings of the International Conference on Nutrition, Dietetics and Sport. Edizioni Minerva Medica, Torino, p 5, 1978
- [Background] Stamler J: Clinical Problems in Hypertension #2. A Patient with Mild Hypertension. A Taped Presentation. Health Learning Systems, Inc, Bloomfield NJ, 1978
- [Background] Stamler J: Epidemiology and Treatment of Hypertension. In: Carlson RJ, Cunningham R, (Eds), Future Directions in Health Care: A New Public Policy, Ballinger Publishing Co, Cambridge, MA, p 95, 1978
- [Background] Stamler J: Population Studies. In: Levy RI, Rifkind BM, Dennis BH, Ernst ND, (Eds), Nutrition, Lipids, and Coronary Heart Disease--A Global View, Raven Press, New York, p 25, 1979
- [Background] Persky VW, Dyer AR, Idris-Soven E, Stamler J, Shekelle RB, Schoenberger JA, Berkson DM, Lindberg HA. Uric acid: a risk factor for coronary heart disease? Circulation. 1979 May;59(5):969-77. doi: 10.1161/01.cir.59.5.969. PMID 428108
- [Background] Persky V, Dyer A, Stamler J, Shekelle RB, Schoenberger J, Wannamaker J, Upton M. The relationship between post-load plasma glucose and blood pressure at different resting heart rates. J Chronic Dis. 1979;32(3):263-8. doi: 10.1016/0021-9681(79)90072-9. No abstract available. PMID 429470
- [Background] Stamler R, Stamler J, Dyer A, Cooper R, Collette P, Berkson DM, Lindberg HA, Stevens E, Schoenberger JA, Shekelle RB, Shekelle S, Paul O, Lepper M, Garside D, Tokich T, Hoeksema R. Asymptomatic hyperglycemia and cardiovascular diseases in three Chicago epidemiologic studies. Diabetes Care. 1979 Mar-Apr;2(2):142-3. doi: 10.2337/diacare.2.2.142. No abstract available. PMID 520117
- [Background] Persky VW, Dyer AR, Stamler J, Shekelle RB, Schoenberger JA. Racial patterns of heart rate in an employed adult population. Am J Epidemiol. 1979 Sep;110(3):274-80. doi: 10.1093/oxfordjournals.aje.a112812. PMID 474564
- [Background] Stamler R, Stamler J, Lindberg HA, Marquardt J, Berkson DM, Paul O, Lepper M, Dyer A, Stevens E. Asymptomatic hyperglycemia and coronary heart disease in middle-aged men in two employed populations in Chicago. J Chronic Dis. 1979;32(11-12):805-15. doi: 10.1016/0021-9681(79)90060-2. No abstract available. PMID 315962
- [Background] Stamler R, Stamler J, Schoenberger JA, Shekelle RB, Collette P, Shekelle S, Dyer A, Garside D, Wannamaker J. Relationship of glucose tolerance to prevalence of ECG abnormalities and to 5-year mortality from cardiovascular disease: findings of the Chicago Heart Association Detection Project in Industry. J Chronic Dis. 1979;32(11-12):817-28. doi: 10.1016/0021-9681(79)90061-4. No abstract available. PMID 315963
- [Background] Joint discussion: the International Collaborative Group. J Chronic Dis. 1979;32(11-12):829-37. No abstract available. PMID 511969
- [Background] Stamler J. Research related to risk factors. Circulation. 1979 Dec;60(7):1575-87. doi: 10.1161/01.cir.60.7.1575. No abstract available. PMID 387286
- [Background] Stamler J: Overweight, Hypertension, Hypercholesterolemia and Coronary Heart Disease. In: Mancini M, (Ed), Medical Complications of Obesity, Proceedings of an International Conference, Naples, Italy, June 1978, Academic Press, London, 191-216, 1979
- [Background] Stamler J: Should Hyperglycemia Always be Treated? In: Mancini M, (Ed), Diet and Drugs in the Treatment of Maturity-Onset Diabetes, Proceedings of a Symposium, Naples, Italy, 28 June 1979
- [Background] Asymptomatic hyperglycemia and coronary heart disease. A series of papers by the International Collaborative Group, based on studies in fifteen populations. Introduction. J Chronic Dis. 1979;32(11-12):683-91. doi: 10.1016/0021-9681(79)90047-x. No abstract available. PMID 315952
- [Background] Stamler J: Hypertension: Aspects of Risk. In: Hunt JC, Cooper T, Frohlich ED, Gifford RW Jr, Kaplan NM, Laragh JH, Maxwell MH, Strong CG (Eds), Hypertension Update: Mechanisms, Epidemiology, Evaluation, Management, Health Learning Systems, Inc, Bloomfield, NJ, pp 23-37, 1979
- [Background] Stamler J. Public health aspects of optimal serum lipid-lipoprotein levels. Prev Med. 1979 Nov;8(6):733-59. doi: 10.1016/0091-7435(79)90357-8. No abstract available. PMID 396531
- [Background] Stamler J: Can An Effective Fat-Modified Diet Be Safely Recommended After Weaning for Infants and Children in General: D. General Discussion. In: Lauer RM, Shekelle RB (Eds), Childhood Prevention of Atherosclerosis and Hypertension, Raven Press, New York, pp 407-410, 1980
- [Background] Dyer AR, Persky V, Stamler J, Paul O, Shekelle RB, Berkson DM, Lepper M, Schoenberger JA, Lindberg HA. Heart rate as a prognostic factor for coronary heart disease and mortality: findings in three Chicago epidemiologic studies. Am J Epidemiol. 1980 Dec;112(6):736-49. doi: 10.1093/oxfordjournals.aje.a113046. PMID 7457467
- [Background] Stamler J: Asymptomatic Hyperglycemia and Risk of Coronary Heart Disease in Middle-Aged Men: American and International Experience. Proceedings, Diabetes and Atherosclerosis Workshop, Dallas, Texas, March 27-29, 1980
- [Background] Stamler J: Data Base on the Major Cardiovascular Diseases in the United States. In: Hegyeli R (Ed), Measurement and Control of Cardiovascular Risk Factors, Atherosclerosis Reviews, Vol. 7, Raven Press, New York, pp 49-96, 1980
- [Background] Stamler J. The established relationship among diet, serum cholesterol and coronary heart disease. Acta Med Scand. 1980;207(6):433-46. doi: 10.1111/j.0954-6820.1980.tb09752.x. No abstract available. PMID 7424562
- [Background] Stamler J. Primary prevention of coronary heart disease: the last 20 years. Am J Cardiol. 1981 Mar;47(3):722-35. No abstract available. PMID 7008572
- [Background] Berkson DM, Stamler J. Epidemiology of the killer chronic diseases. Curr Concepts Nutr. 1981;10:17-55. No abstract available. PMID 7018842
- [Background] Persky V, Dyer AR, Leonas J, Stamler J, Berkson DM, Lindberg HA, Paul O, Shekelle RB, Lepper MH, Schoenberger JA. Heart rate: a risk factor for cancer? Am J Epidemiol. 1981 Oct;114(4):477-87. doi: 10.1093/oxfordjournals.aje.a113213. PMID 7304578
- [Background] Dyer AR, Stamler J, Paul O, Shekelle RB, Schoenberger JA, Berkson DM, Lepper M, Collette P, Shekelle S, Lindberg HA. Serum cholesterol and risk of death from cancer and other causes in three Chicago epidemiological studies. J Chronic Dis. 1981;34(6):249-60. doi: 10.1016/0021-9681(81)90030-8. No abstract available. PMID 7240364
- [Background] Stamler J: Improved Life Styles: Their Potential for the Primary Prevention of Atherosclerosis and Hypertension in Childhood. In: Childhood Prevention of Atherosclerosis and Hypertension, Raven Press, New York, 1980
- [Background] Stamler J, Stamler R: Maturity-Onset Diabetes and Asymptomatic Hyperglycemia. Diabetes and Atherosclerosis Workshop, Sponsored by the Juvenile Diabetes Foundation and the National Heart, Lung, and Blood Institute, Dallas TX, March 27-29, 1980, Juvenile Diabetes Foundation, New York, pp 17-43, 1981
- [Background] Cedres BL, Liu K, Stamler J, Dyer AR, Stamler R, Berkson DM, Paul O, Lepper M, Lindberg HA, Marquardt J, Stevens E, Schoenberger JA, Shekelle RB, Collette P, Garside D. Independent contribution of electrocardiographic abnormalities to risk of death from coronary heart disease, cardiovascular diseases and all causes. Findings of three Chicago epidemiologic studies. Circulation. 1982 Jan;65(1):146-53. doi: 10.1161/01.cir.65.1.146. No abstract available. PMID 7053275
- [Background] Shekelle RB, Paul O, Shryock AM, Stamler J: Dietary Lipids, Serum Cholesterol Concentration, and Risk of Death from Coronary Heart Disease. In: Noseda G, Fragiacomo C, Fumagalli R, Paoletti R (Eds). Lipoproteins and Coronary Atherosclerosis, Elsevier Biomedical Press BV, Amsterdam, pp 87-94, 1982
- [Background] Dyer AR, Stamler J, Shekelle RB, Schoenberger JA, Stamler R, Shekelle S, Berkson DM, Paul O, Lepper MH, Lindberg HA. Pulse pressure-I. Level and associated factors in four Chicago epidemiologic studies. J Chronic Dis. 1982;35(4):259-73. doi: 10.1016/0021-9681(82)90082-0. PMID 7061682
- [Background] Dyer AR, Stamler J, Shekelle RB, Schoenberger JA, Stamler R, Shekelle S, Berkson DM, Paul O, Lepper MH, Lindberg HA. Pulse pressure-II. Factors associated with follow-up values in three Chicago epidemiologic studies. J Chronic Dis. 1982;35(4):275-82. doi: 10.1016/0021-9681(82)90083-2. PMID 7061683
- [Background] Dyer AR, Stamler J, Shekelle RB, Schoenberger JA, Stamler R, Shekelle S, Collette P, Berkson DM, Paul O, Lepper MH, Lindberg HA. Pulse pressure-III. Prognostic significance in four Chicago epidemiologic studies. J Chronic Dis. 1982;35(4):283-94. doi: 10.1016/0021-9681(82)90084-4. PMID 7061684
- [Background] Shekelle RB, Stamler J, Paul O, Shryock AM, Liu S, Lepper M. Dietary lipids and serum cholesterol level: change in diet confounds the cross-sectional association. Am J Epidemiol. 1982 Apr;115(4):506-14. doi: 10.1093/oxfordjournals.aje.a113332. PMID 7041632
- [Background] Orencia AJ, Daviglus ML, Dyer AR, Walsh M, Greenland P, Stamler J. One-hour postload plasma glucose and risks of fatal coronary heart disease and stroke among nondiabetic men and women: the Chicago Heart Association Detection Project in Industry (CHA) Study. J Clin Epidemiol. 1997 Dec;50(12):1369-76. doi: 10.1016/s0895-4356(97)00201-1. PMID 9449940
- [Background] Daviglus ML, Orencia AJ, Dyer AR, Liu K, Morris DK, Persky V, Chavez N, Goldberg J, Drum M, Shekelle RB, Stamler J. Dietary vitamin C, beta-carotene and 30-year risk of stroke: results from the Western Electric Study. Neuroepidemiology. 1997;16(2):69-77. doi: 10.1159/000109673. PMID 9057168
- [Background] Daviglus ML, Dyer AR, Persky V, Chavez N, Drum M, Goldberg J, Liu K, Morris DK, Shekelle RB, Stamler J. Dietary beta-carotene, vitamin C, and risk of prostate cancer: results from the Western Electric Study. Epidemiology. 1996 Sep;7(5):472-7. PMID 8862976
- [Background] Spataro JA, Dyer AR, Stamler J, Shekelle RB, Greenlund K, Garside D. Measures of adiposity and coronary heart disease mortality in the Chicago Western Electric Company Study. J Clin Epidemiol. 1996 Aug;49(8):849-57. doi: 10.1016/0895-4356(96)00067-4. PMID 8699203
- [Background] Lowe LP, Liu K, Greenland P, Metzger BE, Dyer AR, Stamler J. Diabetes, asymptomatic hyperglycemia, and 22-year mortality in black and white men. The Chicago Heart Association Detection Project in Industry Study. Diabetes Care. 1997 Feb;20(2):163-9. doi: 10.2337/diacare.20.2.163. PMID 9118765
- [Background] Greenland P, Daviglus ML, Dyer AR, Liu K, Huang CF, Goldberger JJ, Stamler J. Resting heart rate is a risk factor for cardiovascular and noncardiovascular mortality: the Chicago Heart Association Detection Project in Industry. Am J Epidemiol. 1999 May 1;149(9):853-62. doi: 10.1093/oxfordjournals.aje.a009901. PMID 10221322
- [Background] Stamler J, Stamler R, Neaton JD, Wentworth D, Daviglus ML, Garside D, Dyer AR, Liu K, Greenland P. Low risk-factor profile and long-term cardiovascular and noncardiovascular mortality and life expectancy: findings for 5 large cohorts of young adult and middle-aged men and women. JAMA. 1999 Dec 1;282(21):2012-8. doi: 10.1001/jama.282.21.2012. PMID 10591383
- [Background] Daviglus ML, Liao Y, Greenland P, Dyer AR, Liu K, Xie X, Huang CF, Prineas RJ, Stamler J. Association of nonspecific minor ST-T abnormalities with cardiovascular mortality: the Chicago Western Electric Study. JAMA. 1999 Feb 10;281(6):530-6. doi: 10.1001/jama.281.6.530. PMID 10022109
- [Background] Lowe LP, Greenland P, Ruth KJ, Dyer AR, Stamler R, Stamler J. Impact of major cardiovascular disease risk factors, particularly in combination, on 22-year mortality in women and men. Arch Intern Med. 1998 Oct 12;158(18):2007-14. doi: 10.1001/archinte.158.18.2007. PMID 9778200
- [Background] Daviglus ML, Liu K, Greenland P, Dyer AR, Garside DB, Manheim L, Lowe LP, Rodin M, Lubitz J, Stamler J. Benefit of a favorable cardiovascular risk-factor profile in middle age with respect to Medicare costs. N Engl J Med. 1998 Oct 15;339(16):1122-9. doi: 10.1056/NEJM199810153391606. PMID 9770560
- [Background] Stamler J, Daviglus ML, Garside DB, Dyer AR, Greenland P, Neaton JD. Relationship of baseline serum cholesterol levels in 3 large cohorts of younger men to long-term coronary, cardiovascular, and all-cause mortality and to longevity. JAMA. 2000 Jul 19;284(3):311-8. doi: 10.1001/jama.284.3.311. PMID 10891962
- [Background] Dyer AR, Stamler J, Greenland P. Associations of weight change and weight variability with cardiovascular and all-cause mortality in the Chicago Western Electric Company Study. Am J Epidemiol. 2000 Aug 15;152(4):324-33. doi: 10.1093/aje/152.4.324. PMID 10968377
- [Background] Navas-Nacher EL, Colangelo L, Beam C, Greenland P. Risk factors for coronary heart disease in men 18 to 39 years of age. Ann Intern Med. 2001 Mar 20;134(6):433-9. doi: 10.7326/0003-4819-134-6-200103200-00007. PMID 11255518
- [Background] Blanco-Cedres L, Daviglus ML, Garside DB, Liu K, Pirzada A, Stamler J, Greenland P. Relation of cigarette smoking to 25-year mortality in middle-aged men with low baseline serum cholesterol: the Chicago Heart Association Detection Project in Industry. Am J Epidemiol. 2002 Feb 15;155(4):354-60. doi: 10.1093/aje/155.4.354. PMID 11836200
- [Background] Gapstur SM, Gann PH, Colangelo LA, Barron-Simpson R, Kopp P, Dyer A, Liu K. Postload plasma glucose concentration and 27-year prostate cancer mortality (United States). Cancer Causes Control. 2001 Oct;12(8):763-72. doi: 10.1023/a:1011279907108. PMID 11562117
- [Background] Miura K, Daviglus ML, Dyer AR, Liu K, Garside DB, Stamler J, Greenland P. Relationship of blood pressure to 25-year mortality due to coronary heart disease, cardiovascular diseases, and all causes in young adult men: the Chicago Heart Association Detection Project in Industry. Arch Intern Med. 2001 Jun 25;161(12):1501-8. doi: 10.1001/archinte.161.12.1501. PMID 11427097
- [Background] Stamler J, Liu K, Ruth KJ, Pryer J, Greenland P. Eight-year blood pressure change in middle-aged men: relationship to multiple nutrients. Hypertension. 2002 May;39(5):1000-6. doi: 10.1161/01.hyp.0000016178.80811.d9. PMID 12019283
- [Background] Miura K, Dyer AR, Greenland P, Daviglus ML, Hill M, Liu K, Garside DB, Stamler J; Chicago Heart Association. Pulse pressure compared with other blood pressure indexes in the prediction of 25-year cardiovascular and all-cause mortality rates: The Chicago Heart Association Detection Project in Industry Study. Hypertension. 2001 Aug;38(2):232-7. doi: 10.1161/01.hyp.38.2.232. PMID 11509482
- [Background] Colangelo LA, Gapstur SM, Gann PH, Dyer AR, Liu K. Colorectal cancer mortality and factors related to the insulin resistance syndrome. Cancer Epidemiol Biomarkers Prev. 2002 Apr;11(4):385-91. PMID 11927499
- [Background] Rodin MB, Daviglus ML, Wong GC, Liu K, Garside DB, Greenland P, Stamler J. Middle age cardiovascular risk factors and abdominal aortic aneurysm in older age. Hypertension. 2003 Jul;42(1):61-8. doi: 10.1161/01.HYP.0000078829.02288.98. Epub 2003 Jun 9. PMID 12796281
- [Background] Greenland P, Xie X, Liu K, Colangelo L, Liao Y, Daviglus ML, Agulnek AN, Stamler J. Impact of minor electrocardiographic ST-segment and/or T-wave abnormalities on cardiovascular mortality during long-term follow-up. Am J Cardiol. 2003 May 1;91(9):1068-74. doi: 10.1016/s0002-9149(03)00150-4. PMID 12714148
- [Background] Colangelo LA, Gapstur SM, Gann PH, Dyer AR. Cigarette smoking and colorectal carcinoma mortality in a cohort with long-term follow-up. Cancer. 2004 Jan 15;100(2):288-93. doi: 10.1002/cncr.11923. PMID 14716762
- [Background] Pirzada A, Yan LL, Garside DB, Schiffer L, Dyer AR, Daviglus ML. Response rates to a questionnaire 26 years after baseline examination with minimal interim participant contact and baseline differences between respondents and nonrespondents. Am J Epidemiol. 2004 Jan 1;159(1):94-101. doi: 10.1093/aje/kwh012. PMID 14693664
- [Background] Greenland P, Knoll MD, Stamler J, Neaton JD, Dyer AR, Garside DB, Wilson PW. Major risk factors as antecedents of fatal and nonfatal coronary heart disease events. JAMA. 2003 Aug 20;290(7):891-7. doi: 10.1001/jama.290.7.891. PMID 12928465
- [Background] Dyer AR, Stamler J, Garside DB, Greenland P. Long-term consequences of body mass index for cardiovascular mortality: the Chicago Heart Association Detection Project in Industry study. Ann Epidemiol. 2004 Feb;14(2):101-8. doi: 10.1016/S1047-2797(03)00121-2. PMID 15018882
- [Background] Daviglus ML, Stamler J, Pirzada A, Yan LL, Garside DB, Liu K, Wang R, Dyer AR, Lloyd-Jones DM, Greenland P. Favorable cardiovascular risk profile in young women and long-term risk of cardiovascular and all-cause mortality. JAMA. 2004 Oct 6;292(13):1588-92. doi: 10.1001/jama.292.13.1588. PMID 15467061
- [Background] Daviglus ML, Pirzada A, Liu K, Yan LL, Garside DB, Dyer AR, Hoff JA, Kondos GT, Greenland P, Stamler J. Comparison of low risk and higher risk profiles in middle age to frequency and quantity of coronary artery calcium years later. Am J Cardiol. 2004 Aug 1;94(3):367-9. doi: 10.1016/j.amjcard.2004.04.038. PMID 15276108
- [Background] Daviglus ML, Liu K, Yan LL, Pirzada A, Manheim L, Manning W, Garside DB, Wang R, Dyer AR, Greenland P, Stamler J. Relation of body mass index in young adulthood and middle age to Medicare expenditures in older age. JAMA. 2004 Dec 8;292(22):2743-9. doi: 10.1001/jama.292.22.2743. PMID 15585734
- [Background] Miura K, Greenland P, Stamler J, Liu K, Daviglus ML, Nakagawa H. Relation of vegetable, fruit, and meat intake to 7-year blood pressure change in middle-aged men: the Chicago Western Electric Study. Am J Epidemiol. 2004 Mar 15;159(6):572-80. doi: 10.1093/aje/kwh085. PMID 15003961
- [Background] Daviglus ML, Liu K, Pirzada A, Yan LL, Garside DB, Greenland P, Manheim LM, Dyer AR, Wang R, Lubitz J, Manning WG, Fries JF, Stamler J. Cardiovascular risk profile earlier in life and Medicare costs in the last year of life. Arch Intern Med. 2005 May 9;165(9):1028-34. doi: 10.1001/archinte.165.9.1028. PMID 15883242
- [Background] Liu K, Dyer AR, Vu TH, Pirzada A, Manheim LM, Manning WG, Ashraf MS, Garside DB, Daviglus ML. One-hour postload plasma glucose in middle age and Medicare expenditures in older age among nondiabetic men and women: the Chicago Heart Association Detection Project in Industry. Diabetes Care. 2005 May;28(5):1057-62. doi: 10.2337/diacare.28.5.1057. PMID 15855567
- [Background] Daviglus ML, Liu K, Pirzada A, Yan LL, Garside DB, Wang R, Van Horn L, Manning WG, Manheim LM, Dyer AR, Greenland P, Stamler J. Relationship of fruit and vegetable consumption in middle-aged men to medicare expenditures in older age: the Chicago Western Electric Study. J Am Diet Assoc. 2005 Nov;105(11):1735-44. doi: 10.1016/j.jada.2005.08.008. PMID 16256757
- [Background] Yan LL, Daviglus ML, Liu K, Stamler J, Wang R, Pirzada A, Garside DB, Dyer AR, Van Horn L, Liao Y, Fries JF, Greenland P. Midlife body mass index and hospitalization and mortality in older age. JAMA. 2006 Jan 11;295(2):190-8. doi: 10.1001/jama.295.2.190. PMID 16403931
- [Background] Shekelle RB, Rossof AH, Stamler J. Dietary cholesterol and incidence of lung cancer: the Western Electric Study. Am J Epidemiol. 1991 Sep 1;134(5):480-4; discussion 543-4. doi: 10.1093/oxfordjournals.aje.a116119. PMID 1845471
- [Background] Daviglus ML, Stamler J, Orencia AJ, Dyer AR, Liu K, Greenland P, Walsh MK, Morris D, Shekelle RB. Fish consumption and the 30-year risk of fatal myocardial infarction. N Engl J Med. 1997 Apr 10;336(15):1046-53. doi: 10.1056/NEJM199704103361502. PMID 9091800